CLINICAL TRIAL: NCT02168868
Title: Proteomic Biomarker Tests in Blood Samples from Children with Autism Spectrum Disorder (ASD)
Status: Recruiting | Type: Observational
Sponsor: Benjamin Gesundheit (Industry)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor-Investigator, Benjamin Gesundheit, CEO, Cell El Ltd
Organization: Cell El Ltd (Industry)
Other Study IDs: CellEL-920130030
Record Dates: First submitted 2014-06-19; First posted 2014-06-20 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2023-02

CONDITIONS: Autistic Disorder
Keywords: Autoimmune Diseases; Child Development Disorders; Inflammation; Risk Factors; Pervasive; Autism; Autistic Disorder
MeSH Terms: conditions — Autistic Disorder; Autoimmune Diseases; Developmental Disabilities; Inflammation | interventions — Blood Specimen Collection; Occult Blood; Urinalysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood, urine and stool samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Control Group of Young Children: 2-12 years old age & sex-matched controls - typically developing (TD) children
  Interventions: Diagnostic Test: Blood draw
- Young Children-Autism Spectrum Disorder: 2-12 years old children diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00)
  Interventions: Diagnostic Test: Blood draw
- Young Children-Autism Spectrum Disorder+SCT: 2-12 years old children diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00) due to undergo stem cell transplantation therapy
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Stool Sample Collection; Diagnostic Test: Urine Sample Collection
- High-risk infants: Infants aged 10-19 months not diagnosed with ASD but with a sibling diagnosed with ASD
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Stool Sample Collection
- Mothers of high-risk infants: Mothers of recruited infants aged 10-19 months not diagnosed with ASD but with a sibling diagnosed with ASD
  Interventions: Diagnostic Test: Blood draw
- Adolescent-Autism Spectrum Disorder+SCT: 12-18 years old children diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00) due to undergo stem cell transplantation therapy
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Stool Sample Collection; Diagnostic Test: Urine Sample Collection

INTERVENTIONS:
Diagnostic Test: Blood draw — A blood sample (5 mL) will be collected.
  Other Names: blood sample; venepuncture
Diagnostic Test: Stool Sample Collection — Subjects will be provided a dry, plastic, screw-top specimen container and will be asked to collect a stool sample at home.
  Other Names: Stool Analysis
  Groups: Adolescent-Autism Spectrum Disorder+SCT; High-risk infants; Young Children-Autism Spectrum Disorder+SCT
Diagnostic Test: Urine Sample Collection — Subjects will be provided a dry, plastic, screw-top specimen container and will be asked to collect a urine sample at home.
  Other Names: Urinalysis
  Groups: Adolescent-Autism Spectrum Disorder+SCT; Young Children-Autism Spectrum Disorder+SCT

SUMMARY:
Behavioral testing is the gold standard for diagnosing autism spectrum disorder (ASD). These tests, including ADOS and ADI-R, are subjective, require trained staff to administer, are time-consuming, and can only be administered at a later age. Blood-, urine- or stool-based diagnostic biomarker test for ASD would enable objective early diagnosis, potentially even before clinical symptoms are present, eliminate the need for trained staff and enable early intervention. Such a test would not only conserve money and time but would also provide clues to ASD pathogenesis.

To date, no definitive treatment exists for ASD. Most therapies are symptom-focused, generally focusing on behavioral, social and communication skills. Recent works have reported on promising outcomes of mesenchymal stem cell (MSC) treatment of children with ASD. MSCs are multipotent, non-hematopoietic, easily isolatable and expandable stem cells involved in tissue repair, immunomodulatory responses and neuromodulation. MSC treatment of children with ASD has reportedly led to improvements in speech, sociability, eye coordination, balance, cognition and overall well-being. At the base of this approach lies the known plasticity of the human brain and immune system in the early childhood years and the ability of MSCs to modulate atypical inflammatory and immune activities. Assessment of ASD biomarker profiles in children with ASD who have undergone one or more SCT sessions may shed light on the mechanism of action, assist in better defining ASD-specific diagnostic markers and monitor treatment outcomes.

DETAILED DESCRIPTION:
There is accumulating evidence that at least a subset of children diagnosed with ASD also have aberrant immune functions. This study will attempt to identify more specifically the nature of the potential immune abnormalities in children.

The study will follow a case-control design, involving the following cohorts:

1. young children (2-12 years) diagnosed with ASD
2. children (12-18 years) diagnosed with ASD
3. age- and sex-matched typically developing children
4. high-risk infants (10-19 months) with at least one sibling with diagnosed ASD
5. mothers of these high-risk infants
6. young children (2-12 years) diagnosed with ASD and scheduled to undergo stem cell transplantation therapy (SCT)

Parents will be asked to complete several questionnaires relating to demographic and anamnestic details and to the child's development.

* A single blood draw from all participants will be performed in the clinic.
* A stool sample will be collected from high-risk infants.
* A stool and urine sample will be collected at home from children due to undergo SCT. For children scheduled to undergo SCT, the blood, stool and urine samples must be collected before therapy.

  * Parents of high-risk infants will be contacted by phone or email when the child reaches diagnosable age (3.5 years) and again at the age of 6 years, to obtain an update on the child's ASD status. If the child has been diagnosed with ASD, an additional blood and stool sample may be collected.
  * Children who underwent SCT will be contacted 2±1 months and 6±1 months after the first treatment session, for collection of additional blood samples. Stool and urine samples will be collected at the 6±1 month post-treatment visit as well. Should the child undergo additional SCT within two years of the first treatment, additional blood, stool and urine samples may be collected. At each subsequent visit, a parent/legal guardian will be asked to complete several short questionnaires.

Adverse events to blood drawing will be reported to the Data Coordinating Center using the appropriate Case Report Form (CRF).

In cases of adverse effects (AE) related to the drawing of blood or performance of examination of patients in the course of standard examination procedures, the investigating team will proceed in accordance with local guidelines (to be inserted by the PI), reporting the incidents which occurred during the course of a clinical trial.

Clinical data will be collected by the investigator, or a person appointed and appropriately trained by the investigator, and shall be entered into standardized CRFs and shared online with the sponsor. Source data will be retained for all data entered in the CRFs. Progress reports and the Final Report at the conclusion of the trial will be submitted to the regulatory authority and the Ethics Committee, as required.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children
2. Child aged 2-12 years with diagnosed ASD according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV (299.00) or DSM-V (299.00) OR Child aged 2-18 years diagnosed ASD according to DSM-IV (299.00) or DSM-V (299.00) AND scheduled to undergo stem cell transplantation OR Child aged 10-19 months not diagnosed with ASD but with a sibling diagnosed with ASD according to (DSM)-IV (299.00) or DSM-V (299.00) (herein termed "high-risk infants") OR Mothers of recruited high-risk infants OR A typically developing child aged 2-12 years with no signs of ASD or history of ASD in the immediate family
3. Informed consent signed by the parent/legal guardian

Exclusion Criteria:

1. Child and/or mother completed treatment with systemic steroids or immune suppressants less than 4 weeks before the screening visit
2. Child and/or mother diagnosed with severe infectious diseases or sepsis over the last 6 months
3. Child with ASD treated for a severe convulsive disorder (intractable seizures)
4. Child and/or mother with hematological or malignant disorder
5. For children in the SCT cohort: No new planned immune-modulating treatment (other than SCT) for at least 6 months before or after planned stem cell transplantation date
6. If the PI suspects that the participant will not comply with study requirements, the participant may be excluded.

Ages: 10 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Up to a total of 350 male and female children, aged 2-12 years, diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00)
  2. Up to a total of 350 male and female typically developing (TD) children aged 2-12 years with no signs of ASD or history of ASD in the immediate family who will serve as controls for the main subset of children with ASD
  3. Up to 50 infants aged 10-19 months not diagnosed with ASD but with a sibling diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00) (herein, high-risk infants)
  4. Up to 50 mothers of the high-risk infants participating in the study
  5. Up to 50 male and female children, aged 2-12 years, diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00) scheduled to undergo stem cell therapy (SCT)
  6. Up to 50 male and female children, aged 12-18 years, diagnosed with ASD according to DSM-IV (299.00) or DSM-V (299.00) scheduled to undergo SCT
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of discriminating proteomic biomarker profile in blood of children with ASD vs. matched TD children | One day
  Finding a proteomic signature in children with ASD
Identification of discriminating proteomic biomarker profiles in blood of high-risk infants, at recruitment vs. after diagnosis of ASD, if diagnosed | Up to 5 years after initial blood draw
  Finding a proteomic signature in infants at high-risk of ASD
Comparison of blood biomarker profiles in ASD children before versus after SCT | Through study completion, up to 6 months
  Finding ASD-specific blood proteomic biomarkers that can be modified by SCT

SECONDARY OUTCOMES:
ASD severity vs. blood biomarker levels | Through study, up to 5 years, depending on cohort
  Correlative assessment of ASD severity vs. blood biomarker levels
Blood biomarker levels and SCT outcomes | Through study completion, up to 6 months
  Correlative assessment of blood biomarker levels and SCT outcomes

OTHER OUTCOMES:
Identification of ASD-specific proteomic biomarkers and/or microbiome profile in stool samples of children with ASD before vs. after SCT | Up to 6 months
  Identification of an ASD-associated proteomic/microbiome signature that may be altered by SCT
Comparison of urine biomarker profiles in ASD children before versus after SCT | Up to 6 months
  Finding ASD-specific urine proteomic biomarkers that can be modified by SCT
Identification of ASD-specific proteomic biomarker and microbiome signature in stool samples of high-risk infants before vs. after ASD diagnosis, if diagnosed | Through study completion, up to 5 years
  Finding proteomic biomarker or microbiome signature in stool samples of high-risk infants that changes after diagnosis of ASD
Identification of discriminating proteomic profiles in blood of the mothers of high-risk infants | One day
  Finding a proteomic signature that can identify mothers at risk of having an ASD child
Correlative assessment of proteomic biomarker expression in the high-risk infant and his/her mother | 1 day
  Comparison of blood proteomic signature of a mother of a high-risk infant vs. that of the high-risk infant

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Gesundheit, MD, Principal Investigator — Cell El Ltd
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Gesundheit B, Rosenzweig JP, Naor D, Lerer B, Zachor DA, Prochazka V, Melamed M, Kristt DA, Steinberg A, Shulman C, Hwang P, Koren G, Walfisch A, Passweg JR, Snowden JA, Tamouza R, Leboyer M, Farge-Bancel D, Ashwood P. Immunological and autoimmune considerations of Autism Spectrum Disorders. J Autoimmun. 2013 Aug;44:1-7. doi: 10.1016/j.jaut.2013.05.005. Epub 2013 Jul 15. PMID 23867105
- [Background] Gesundheit B, Zisman PD, Hochbaum L, Posen Y, Steinberg A, Friedman G, Ravkin HD, Rubin E, Faktor O, Ellis R. Autism spectrum disorder diagnosis using a new panel of immune- and inflammatory-related serum biomarkers: A case-control multicenter study. Front Pediatr. 2023 Feb 21;11:967954. doi: 10.3389/fped.2023.967954. eCollection 2023. PMID 36896401